CLINICAL TRIAL: NCT07030803
Title: Comparative Study of the Efficacy of Treatment of Idiopathic Overactive Bladder (OAB) in Children: Oxybutynine vs. Transcutaneous Neurostimulation
Acronym: HAV-O-TENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2023_843_0176
Record Dates: First submitted 2025-04-29; First posted 2025-06-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Overactive Bladder (OAB); Transcutaneous Neurostimulation; Posterior Tibial Nerve Stimulation
Keywords: Overactive Bladder; transcutaneous neurostimulation; posterior tibial nerve stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxybutynin (Active Comparator)
  Interventions: Other: Oxybutynin
- TENS (Experimental)
  Interventions: Device: medical device Urostim

INTERVENTIONS:
Other: Oxybutynin — oxybutynin
  Arms: oxybutynin
Device: medical device Urostim — medical device used to deliver posterior tibial nerve stimulation (PTNS)
  Arms: TENS

SUMMARY:
The absence of infectious, urological and neurological causes defines the idiopathic character of overactive bladder (OAB). Although a progressive approach starting with behavioural therapy (urotherapy) is recommended, anticholinergic agents remain the mainstay of medical treatment of overactive bladder (OAB) in children. Bladder neuromodulation is also used but no study with sufficient evidence has assessed its effectiveness and tolerance compared to the reference treatment. The purpose of HAV-O-TENS is to demonstrate the non-inferiority of treating idiopathic overactive bladder (OAB) in children using posterior tibial nerve stimulation (PTNS) compared to the reference treatment with oxybutynin after three months of treatment.

Before inclusion, patients will receive instructions for urotherapy and a treatment plan. After confirming the diagnosis and obtaining informed consent, patients will be randomly assigned to either oxybutynin or PTNS (posterior tibial nerve stimulation) treatment, and their effectiveness, tolerance, and adherence will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6 to 16 years
* Showing signs of OAB (pollakiuria (> 8 micturitions/d and/or urgenturia(>x2/week) and/or daytime urine leakage (1/d) and/or nocturia x2/night)
* No treatment for more than 3 months
* Urotherapy rules followed for at least 1 month
* Beneficiary of a social security plan
* Signature of consent by parents/legal guardian(s) and child's agreement

Exclusion Criteria:

* Neurological cause of bladder dysfunction,
* History of pelvic surgery,
* Significant post-micturition residual (> 10% of micturition),
* Recurrent urinary tract infections (> 3) in the 6 months prior to inclusion or urinary tract infection at inclusion.
* Pregnant or breast-feeding adolescents
* Severe constipation resistant to treatment (Rome IV),
* Contraindication to oxybutynin
* Contraindication to the use of TENS (Urostim)

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Variation of DVISS score between PTNS treatment group and oxybutynin group | at 3 months
  DVISS score is : Dysfunctional Voiding and Incontinence Symptoms Score (DVISS) Questionnaire.
  The DVISS is a 13-item instrument that includes 1 QOL question. The first 5 questions are scored using an ordinal scale with the remainder in binary format.
  The DVISS scores are based on the estimated odds ratio (OR) for each question between cases and controls. For example, a score of 1 is given if the item's OR is between 2 and 10, and a score of 5 is given if the OR is greater than 50. The total score can range from 0 to 35 with a cutoff score of 8.5 having 90% sensitivity and specificity at detecting BBD.

SECONDARY OUTCOMES:
variation of treatment duration between both groups | at 6 months
variation of time to treatment efficacy between both groups | at 6 months
variation of tolerance between both groups | at 3 months
variation of tolerance between both groups | at 6 months
variation of compliance between both groups | at 3 months
  variation of compliance between both groups
variation of compliance between both groups | at 6 months
  variation of compliance between both groups
variation of long-term efficacy between both groups | at 12 months
variation of long-term efficacy between both groups | at 18 months
variation of long-term efficacy of AOB frequency between both groups | at 24 months
  Long term efficacy of OAB frequency is measured with DVISS score. The DVISS is a 13-item instrument that includes 1 QOL question. The first 5 questions are scored using an ordinal scale with the remainder in binary format.
  The DVISS scores are based on the estimated odds ratio (OR) for each question between cases and controls. For example, a score of 1 is given if the item's OR is between 2 and 10, and a score of 5 is given if the OR is greater than 50. The total score can range from 0 to 35 with a cutoff score of 8.5 having 90% sensitivity and specificity at detecting BBD.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No